CLINICAL TRIAL: NCT04955496
Title: Evaluation of the Effect of Enhanced Recovery After Surgery for Cervical Surgery
Brief Title: ERAS on Cervical Surgery
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2019195
Record Dates: First submitted 2021-07-01; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Cervical Spondylosis
Keywords: Enhanced Recovery after Surgery, Cervical Spondylosis, Outcome measures
MeSH Terms: conditions — Spondylosis | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERAS Group: Patients were treated by enhanced recovery after surgery
  Interventions: Procedure: Enhanced recovery after surgery
- Control Group: Patients were not treated by enhanced recovery after surgery

INTERVENTIONS:
Procedure: Enhanced recovery after surgery — ERAS management includes 3 parts: (1) Preoperative analgesia and airway evaluation. (2) The protection and reconstruction of the musculo-ligamentous complex during the surgery, the safe intubation, and the local infiltration anesthesia during surgery. (3) Collar free, multimodal analgesia, airway management, and early recovery after surgery.
  Groups: ERAS Group

SUMMARY:
This study is to evaluate the application effect of the concept of accelerated rehabilitation surgery in the perioperative period of patients with cervical spondylosis through a retrospective cohort study

DETAILED DESCRIPTION:
To evaluate the effect of a series of optimization measures in ERAS among the patients during perioperative period who underwent cervical surgery.

Methods:

A retrospective cohort study was conducted for the patients who underwent cervical spine surgery in a top three hospital in Beijing from April to December 2018. According to whether to implement enhanced recovery surgery, the patients were divided into enhanced recovery surgery group (eras group) and control group. The self-designed data collection table was used to collect data in the patient's medical records, including general demographic data and disease treatment data, implementation of accelerated rehabilitation surgery and application effect. Among them, the application effect includes the operation related complications, the visual analog scale (VAS) score of neck and shoulder pain, the ability of daily living after discharge, the length of stay, the cost of hospitalization and other recent rehabilitation effect indicators, as well as the rehospitalization rate of 90 days and the Japanese Orthopaedic Society four months after operation Association (JOA) score, neck disability index (NDI) score, neck and shoulder pain symptoms, neck and shoulder stiffness symptoms and other long-term rehabilitation indicators. Independent sample t-test, rank sum test and chi square test were used to compare the differences between the two groups. On the basis of single factor analysis, combined with multi factor analysis, the impact of groups on outcome indicators was clarified, included 90-day readmission, reexamination time, follow-up JOA score, NDI score, neck and shoulder pain symptoms and neck and shoulder stiffness symptoms.

ELIGIBILITY:
Inclusion Criteria:

* ① patients with cervical spondylosis were definitely diagnosed; ② Cervical spine surgery was performed under general anesthesia; ③ Age ≥ 18 years old;

Exclusion Criteria:

* ① patients with cervical deformity correction surgery; ② Patients who underwent secondary cervical spine surgery; ③ Patients with spinal cord injury caused by trauma (4) patients with thoracic and atlantoaxial diseases and corresponding surgery; ⑤ Ankylosing spondylitis patients; ⑥ Patients with cerebral infarction, cerebral palsy and nerve root injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients who underwent cervical spine surgery
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
the ability of daily living | Baseline
  The medical history related to the ability of daily living
the ability of daily living | 90-day follow-up after surgery
  The medical history related to the ability of daily living
the length of hospital stay | Admission to discharge, an average of 3 days
  the length of hospital stay
the cost of hospitalization | Admission to discharge, an average of 3 days
  the cost of hospitalization
the rehospitalization rate | 90-day follow-up after surgery
  the rehospitalization rate of 90 days

SECONDARY OUTCOMES:
VAS (visual analog scale ) score | Baseline
  VAS score of neck and shoulder pain, 0-100 points, higher means worse outcomes
VAS (visual analog scale ) score | 90-day follow-up after surgery
  VAS score of neck and shoulder pain, 0-100 points, higher means worse outcomes
NDI (neck disability index) score | Baseline
  NDI score, 0-100%, higher means worse outcomes
NDI (neck disability index) score | 90-day follow-up after surgery
  NDI score, 0-100%, higher means worse outcomes
symptoms of neck and shoulder | Baseline
  The presence or absence of neck and shoulder pain symptoms
symptoms of neck and shoulder | 90-day follow-up after surgery
  The presence or absence of neck and shoulder pain symptoms
symptoms of neck and shoulder | Baseline
  The presence or absence of neck and shoulder stiffness symptoms
symptoms of neck and shoulder | 90-day follow-up after surgery
  The presence or absence of neck and shoulder stiffness symptoms
neurological function | Baseline
  the Japanese Orthopaedic Society Association (JOA) score, 0-17 points, lower means worse outcomes
neurological function | 90-day follow-up after surgery
  the Japanese Orthopaedic Society Association (JOA) score, 0-17 points, lower means worse outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No